CLINICAL TRIAL: NCT00102648
Title: Phase I/Ib Study of Sarasar and Temodar in Patients with Recurrent or Temodar-Refractory Glioblastoma Multiforme
Brief Title: Lonafarnib and Temozolomide in Treating Patients with Glioblastoma Multiforme That is Recurrent or Did Not Respond to Previous Treatment with Temozolomide
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 2004-0424; NCI-2012-01311 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2010-00417; 2004-0424 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2005-01-31; First posted 2005-02-01 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Malignant Supratentorial Neoplasm; Recurrent Glioblastoma; Recurrent Gliosarcoma
MeSH Terms: conditions — Supratentorial Neoplasms; Glioblastoma; Gliosarcoma | interventions — lonafarnib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (temozolomide and lonafarnib) (Experimental): Patients receive temozolomide PO QD on days 1-7 and 15-21 and lonafarnib PO BID on days 8-14 and 22-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Lonafarnib; Drug: Temozolomide

INTERVENTIONS:
Drug: Lonafarnib — Given PO
  Other Names: 4-[2-[4-[(11R)-3,10-Dibromo-8-chloro-6,11-dihydro-5H-benzo[5,6]cyclohepta[1,2-b]pyridin-11-yl]-1-piperidinyl]-2-oxoethyl]-1-piperidinecarboxamide; Sarasar; SCH 66336; SCH-66336; SCH66336
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac

SUMMARY:
This phase I trial studies the side effects and best dose of lonafarnib when given together with temozolomide and to see how well they work in treating patients with glioblastoma multiforme that is has come back or did not respond to previous treatment with temozolomide. Lonafarnib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving lonafarnib together with temozolomide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose Sarasar (SCH66336, lonafarnib) when combined with Temodar (temozolomide) in an alternating week schedule.

II. To describe the toxicities of the Sarasar and Temodar combination treatment using this dosing schedule.

III. To evaluate response as measured by 6-month progression-free survival and objective tumor response.

OUTLINE: This is a dose-escalation study of lonafarnib.

Patients receive temozolomide orally (PO) once daily (QD) on days 1-7 and 15-21 and lonafarnib PO twice daily (BID) on days 8-14 and 22-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven supratentorial glioblastoma multiforme (GBM) or gliosarcoma
* Patients must have shown unequivocal evidence for tumor recurrence or progression by magnetic resonance imaging (MRI) scan after radiation therapy; the scan done prior to study entry documenting progression will be reviewed by the treating physician to document tumor volume changes to provide a gross assessment of growth rate
* Patients may have had as many as 2 prior chemotherapy regimens for recurrent or progressive tumor; patients must have had prior treatment with Temodar but may not have had prior treatment with farnesyl transferase inhibitors (Sarasar or Zarnestra); patients in phase 1b expansion are required to have received a minimum of two cycles of adjuvant temozolomide (TMZ)
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of this hospital
* Patients must have shown unequivocal evidence for tumor progression by MRI or computed tomography (CT) scan; a scan should be performed within 14 days prior to registration and on a steroid dose that has been stable or decreasing for at least 5 days; if the steroid dose is increased between the date of imaging and registration a new baseline magnetic resonance (MR)/CT is required; the same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement
* Patients (pts) having had recent resection of recurrent or progressive tumor are eligible as long as:

  * Patients must be status post surgical resection at least 2 weeks prior to study enrollment, have recovered from surgery, have adequate early wound healing and a Karnofsky performance status of > or = 60
  * Residual disease following resection of recurrent tumor is not mandated for eligibility into the study; a CT/MRI should be done within 96 hours (hrs) post-op or at least 4 weeks (wks) post-op (within 14 days of registration); if the steroid dose is increased between the scan date and registration, a new baseline MRI/CT is required on a stable steroid dose for 5 days
* Patients must have a Karnofsky performance status of >= 60
* Patients must have recovered from the toxic effects of prior therapy: 4 weeks from prior cytotoxic therapy and/or at least two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count); any questions related to the definition of non-cytotoxic agents should be directed to the study chair
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count of >= 100,000/mm^3
* Serum glutamic pyruvate transaminase (SGPT) < 2.5 times normal
* Alkaline phosphatase < 2.5 times normal
* Bilirubin < 1.5 mg
* Blood urea nitrogen (BUN) < 1.5 times institutional normal
* Creatinine < 1.5 times institutional normal

Exclusion Criteria:

* Patients must not be taking primidone, carbamazepine, phenobarbital or phenytoin anticonvulsants; patients changing from these anticonvulsants to other allowable drugs that are not enzyme inducing antiepileptic drugs (EIAEDs) must be off the drugs listed above for at least 72 hours prior the initiation of treatment
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), are ineligible unless in complete remission and off of all therapy for that disease for a minimum of 3 years
* Patients must not have:

  * Uncontrolled active infection
  * Disease that will obscure toxicity or dangerously alter drug metabolism
  * Serious intercurrent medical illness
  * Prior recurrence with a farnesyl transferase inhibitor
  * Oral contraceptives and other hormonal methods (Depo-Provera) of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2004-12-21 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of lonafarnib when given with temozolomide, defined as the dose at which fewer than one-third of patients experience dose-limiting toxicity (DLT) | 28 days
Tolerability of regimen in patients with disease progression or recurrence during or after recent completion of treatment with temozolomide | Up to 11 years

SECONDARY OUTCOMES:
Progression free survival (PFS) | 6 months
  In the historical dataset, the proportion of patients remaining alive and free from progression at 6 months was 15% (95% confidence interval for ranged from 10% to 19%). We will set p0 to 15% and we will set p1 to 30% (looking for a doubling of the 6-month PFS rate). Based on these design parameters, a two-stage design would require that at least 4 of the initial 19 patients are without progression at 6 months.
Objective response | Up to 11 years
Overall survival | Up to 11 years
Treatment-related toxicities | Up to 11 years
  Treatment-related toxicity data will be collected and described.

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Puduvalli, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org